CLINICAL TRIAL: NCT00269139
Title: Study of Outcome With an Intervention From the Cape Cod Model of Psychotherapy for Subjects in a Behavioral Crisis and With the Diagnosis of Borderline Personality Disorder (BPD) or Post-Traumatic Stress Disorder (PTSD)
Brief Title: Outcome of Crisis Intervention for Subjects With Borderline Personality Disorder or Post-Traumatic Stress Disorder
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laddis, Andreas, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 719371
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2006-02-20 (Estimated); Status verified 2005-12

CONDITIONS: Borderline Personality Disorder; Post-Traumatic Stress Disorders
Keywords: Behavioral crisis; Perception of social crisis; Repetition compulsion; Intrusive mental events; Uncontrollable urges
MeSH Terms: conditions — Borderline Personality Disorder; Stress Disorders, Post-Traumatic

INTERVENTIONS:
Behavioral: Crisis resolution

SUMMARY:
Dr. Laddis will test a hypothesis about the nature and the management of behavioral crises in patients with borderline personality disorder (BPD) or post-traumatic stress disorder (PTSD). The term "behavioral crisis" is used strictly for periods of uncontrollable urges to repeat mental or outward activity, e.g., flashbacks, cutting, binging on food, drugs or sex, with no intervals to rethink one's priorities or to consider others' direction.

The clinical hypothesis states, in two steps, that:

1. the perception of a life crisis precedes and then underlies every behavioral crisis;
2. the behavioral crisis resolves promptly and all symptoms end if the clinicians engage the patient about his management of the life crisis that underlies the symptoms.

DETAILED DESCRIPTION:
Subjects in the experimental group will be treated by Dr. Laddis after their admission to a crisis stabilization unit (CSU) or to an inpatient unit (IPU) for a behavioral crisis. Subjects will be included at random, as assigned to Dr. Laddis according to his routine duties at those units.

Subjects in the control group will receive treatment for behavioral crisis according to the preference of the clinical staff at other comparable units. That treatment will constitute "treatment as usual". Clinicians in the control settings will not be informed about the experimental hypothesis, the clinical intervention and the contingent outcomes.

The subjects will be tested for the results of treatment 12-24 hours after composition of a treatment plan. The testing will be done with the Brief Psychiatric Rating Scale (BPRS), as well as with a set of criteria devised by Dr. Laddis to measure the outward behavior and the mental events during behavioral crisis. The patients and the attending frontline staff will be interviewed also about their beliefs in regard to what, among the clinicians' interventions, made a difference for the course of the behavioral crisis, for better or for worse. The raters will be trained for interrater reliability and they will not be informed about the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with BPD or PTSD, with a structured interview according to the current diagnostic manual
* In behavioral crisis

Exclusion Criteria:

* Brain damage
* Currently intoxicated with alcohol or drugs or in withdrawal

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) scores
Scores on Client Observation and Client Interview, tools designed for this study

SECONDARY OUTCOMES:
Patient interview and ratings for the value of the clinicians' interventions
Staff interview and ratings for their own interventions

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Laddis, MD, Principal Investigator — Cape Cod and Islands Community Mental Health Center
Locations (1):
- Cape Cod and Islands Community Mental Health Center, Pocasset, Massachusetts, United States

REFERENCES:
- [Derived] Laddis A. Outcome of crisis intervention for borderline personality disorder and post traumatic stress disorder: a model for modification of the mechanism of disorder in complex post traumatic syndromes. Ann Gen Psychiatry. 2010 Apr 27;9:19. doi: 10.1186/1744-859X-9-19. PMID 20420716